CLINICAL TRIAL: NCT00886925
Title: Effects of the Administration of Albumin in Patients With Cirrhosis and Acute Hepatic Encephalopathy.
Brief Title: Efficacy of Albumin for Acute Encephalopathy in Patients With Cirrhosis
Acronym: ALFAE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALFAE; 2008-003376-21 (EudraCT Number); PI07 - 0641 (Other Grant/Funding Number: FIS (Instituto de Salud Carlos III))
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-04

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic encephalopathy; Cirrhosis; Albumin
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Albumins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albumin (Active Comparator)
  Interventions: Drug: Albumin
- Saline (Placebo Comparator)
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Albumin — Albumin 20%. Day 0: 400-600 ml. Day 2: 200-400 ml.
  Arms: Albumin
Drug: Sodium chloride 0.9% — Day 0: 400-600 ml. Day 2: 200-400 ml.
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether the administration of albumin in addition to the standard care is effective in the treatment of an episode of hepatic encephalopathy in patients with cirrhosis.

DETAILED DESCRIPTION:
Hepatic encephalopathy is a frequent complication of cirrhosis that is usually associated with poor prognosis. The most common presentation is an acute episode of hepatic encephalopathy precipitated by factors that increase the exposure of the brain to ammonia. Current therapies are based on measures that decrease plasma ammonia and counteract the effect of factors such as infection or electrolyte's disturbances. Brain edema and abnormalities of cerebral blood flow appear to be important. Part of the impairment of astrocyte function could be related to an increase of oxidative stress injury.

In patients with cirrhosis and hepatic encephalopathy, the concentration of albumin in plasma is usually low. Administration of human albumin in patients with hepatorenal syndrome and spontaneous bacterial peritonitis has a major impact on the prognosis of these complications. Albumin prevents circulatory dysfunction and renal failure. The mechanisms of action may include the maintenance of oncotic pressure and a scavenger effect of toxic substances present in blood. Albumin has also shown beneficial effects in neurological injury secondary to stroke, probably in relation to this scavenger effect.

The administration of intravenous albumin to patients with hepatic encephalopathy may have beneficial effects on the course of encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis of the liver
* Hepatic encephalopathy stage>1
* Completion of a standardized protocol to investigate precipitating factors
* Informed consent by next of keen

Exclusion Criteria:

* Pregnancy
* Terminal liver disease (advanced liver disease and performance status 3-4 prior to the episode of acute encephalopathy)
* Need of advanced life support (mechanical ventilation, ionotropic support, dialysis)
* Need of albumin administration (e.g. bacterial spontaneous peritonitis)
* Contraindication for albumin administration (e.g. cardiac failure)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without hepatic encephalopathy | Day 3

SECONDARY OUTCOMES:
Severity of encephalopathy assessed by CHESS and West-Haven | Admission to the hospital (up to day 14)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Cordoba, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (4):
- Spain (4):
  - Parc Tauli, Sabadell, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic, Barcelona

REFERENCES:
- [Derived] Simon-Talero M, Garcia-Martinez R, Torrens M, Augustin S, Gomez S, Pereira G, Guevara M, Gines P, Soriano G, Roman E, Sanchez-Delgado J, Ferrer R, Nieto JC, Sunye P, Fuentes I, Esteban R, Cordoba J. Effects of intravenous albumin in patients with cirrhosis and episodic hepatic encephalopathy: a randomized double-blind study. J Hepatol. 2013 Dec;59(6):1184-92. doi: 10.1016/j.jhep.2013.07.020. Epub 2013 Jul 19. PMID 23872605